CLINICAL TRIAL: NCT05487937
Title: Evaluation of Toleriane Ultra Reno in Allergic Subjects Having Skin Intolerance to Their Usual Cosmetic Care for One Month
Brief Title: Toleriane Ultra Reno in Allergic Subjects With Skin Intolerance to Their Usual Cosmetic
Status: Completed | Type: Observational
Sponsor: Cosmetique Active International (Industry)
Responsible Party: Sponsor
Other Study IDs: LRP20006-TOLERIANE ULTRA
Record Dates: First submitted 2022-06-17; First posted 2022-08-04 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Allergy
Keywords: allergy; intolerance; dermocosmetic; allergic
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Toleriane Ultra: Participants are asked to apply the study product twice daily (morning and evening) at home for 28 days.
  Interventions: Other: Use of Toleriane Ultra to relieve face allergic skin

INTERVENTIONS:
Other: Use of Toleriane Ultra to relieve face allergic skin — The product developed to restore the natural skin barrier and rebalance skin immune system is a white cream and is applied on the face by a slight massage under normal conditions of use twice daily for 28 days.

SUMMARY:
Sensitive skin is a subjective cutaneous hyper-reactivity to environmental factors. People report exaggerated reactions when their skin, especially on the face, is in contact with substances such as cosmetics. For this reason, Toleriane Ultra has been developed to limit the risk of allergy and relieve skin discomfort. The study aims at demonstrating that Toleriane Ultra is well tolerated in participants with allergic background and having experienced former intolerance to their cosmetic or toiletries routine, and improves skin sensitivity in such individuals.

This open-labeled, multicenter study was conducted under dermatological control in Caucasian subjects above 16 years of age with an allergic background and intolerance to cosmetics lasting for at least 2 years prior to inclusion. The dermocosmetic product was to be applied on the entire face twice daily for 28 days.

DETAILED DESCRIPTION:
The evaluation of Toleriane Ultra in allergic subjects having skin intolerance to their usual cosmetic care has been conducted under cosmetic form and dermatological control by Dermscan that is certified by the International Standards Organization (ISO) 9001-2015.

Each study report is subjected to a quality inspection by a member of Dermscan. A certificate of quality inspection signed by a proofreader (not involved in the audited study) is enclosed in each study. The inspection of the study report allows to confirm that the results reflect exactly the study raw data and that the study fulfills any standard and regulatory requirements.

With regard to the statistical analysis, the continuous data is summarized using the following statistics by time point (Day0, Day14, Day28): number of values, mean, median, standard deviation, minimum value, maximum value. For each continuous data obtained from devices (Tewameter for Transepidermal water loss, Corneometer for cutaneous hydration measurements), a mixed linear model for repeated measurements is adjusted to raw data, including the factor "time" as fixed (with 3 levels: Day0, Day14, Day28) and the factor "subject" as random. Using the adjusted means obtained from this model (LS-Means), the contrast of interest is built to assess the change from baseline (Day0) at each point (Day14 and D28). For the categorical data, the global tolerance scores by both the investigator and the participant assessed using a 4-point scale are summarized in frequency (N) and percentage (%) by time point (Day14, D28) with associated 95% confidential interval. For other categorical data, a Wilcoxon signed rank test is carried out for each parameter assessed using an ordinal scale:

* Sensiscore (erythema, irritation, stinging, itching, burning, tightening, discomfort) assessed using a 5-point structured scale of frequency and intensity of the functional signs.
* Composite score of the skin state (redness, pruritus, dryness, burning sensation, tingling) assessed using a 4-point structured scale.
* Smoothing effect assessed using a 4-point structured scale.

The participants have the right to exit from the study at any time and for any motive, in compliance with the Helsinki Declaration (1964) and its successive updates. The investigator can also interrupt the person's participation in the study prematurely in the case of a disease occurrence, a pregnancy or the occurrence of an adverse reaction.

Every premature exit must be classified under one of the following headings:

* presence of non-inclusion criteria;
* Undesirable Effect / Adverse Event occurrence;
* Serious Adverse Event / Serious Adverse Effect occurrence;
* withdrawal of consent;
* lost to follow-up;
* the appearance of non-inclusion criteria;
* non-adherence to the protocol;
* other reason.

All the adverse events and serious adverse events are reported in the case report form and the study report.

No replacement is foreseen as 10% additional participants are planned to be included in the study (110 included participants in order to obtain results on 100 (+/- 10%) participants minimum.). An identification code is attributed to each participant for the purpose to keep his/her identity confidential.

The personnel in charge of the study collects data into individual case report forms in electronic or paper format and/or directly from measurement software. When information is collected in paper format, the double data entry is then done from these supports by the designed operator(s), without any interpretation, in specific EXCEL databases. The Project Manager or assistant checks the double data entry by comparing both databases. Then the coherence of the whole data set is checked as well as formulas used in the EXCEL tables (calculation formulas, selected data…). When all the controls are done, the database is locked.

ELIGIBILITY:
Inclusion Criteria:

* 16 years old and above
* caucasian
* phototype I to IV
* participants presenting with an allergy ground
* participants without visible allergic dermatosis at inclusion on the face
* participants having skin intolerance with cosmetic care
* participants who have not changed their cosmetic habits for less than 15 days

Exclusion Criteria:

* for women: pregnant or nursing or planning a pregnancy during the study
* cutaneous pathology on the studied zone
* use of topical or systemic treatment during the previous weeks liable to interfere with assessment of the cutaneous acceptability of the study product
* professional facial care during the study or within the previous month
* excessive exposure to sunlight or UV-rays within the previous month
* participant having undergone surgery under general anesthesia within the previous month

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: participants meeting the inclusion and exclusion criteria and accepting the study constraints
Sampling Method: Non-Probability Sample
Enrollment: 109 (Actual)
Dates: Start 2021-05-25 (Actual); Primary Completion 2021-09-28 (Actual); Study Completion 2021-09-28 (Actual)

PRIMARY OUTCOMES:
change in cutaneous acceptability | Change from baseline to Day28
  evaluation of global tolerance by investigator and participants on a 4-point scale
change in cutaneous reactivity score | Change from baseline to Day28
  cutaneous reactivity score on a 4-point scale (non stinging, mild stinging sensation, moderate stinging sensation, severe stinging sensation) before and after product use with a stinging test
change in Sensiscore | Change from baseline to Day28
  questionnaire on frequency and intensity of functional signs on the face by self-assessment on a 5-point scale
change in composite score | Change from baseline to Day28
  questionnaire on pruritus, redness, burning and tingling by self-assessment on a 4-point scale
change in transepidermal water loss | Change from baseline to Day28
  transepidermal water loss measurements before and after product use with a Tewameter
change in the hydration rate | Change from baseline to Day28
  hydration rate before and after product use with a Corneometer

CONTACTS AND LOCATIONS:
Overall Officials: Anna Czermanska, Study Director
Locations (1):
- Dermscan Poland Sp. z o. o., Gdansk, Poland

REFERENCES:
- [Derived] Kerob D, Czermanska A, Karamon EM, Moga A, Lecerf G, Niore M, Le Dantec G, Le Floc'h C, Tan J. A Dermocosmetic Significantly Reduces the Frequency and Intensity of Facial Skin Intolerability and Sensitivity in Subjects with Skin Intolerant to Skin Care Products and Sensitive Skin. Clin Cosmet Investig Dermatol. 2023 Jul 11;16:1787-1794. doi: 10.2147/CCID.S418483. eCollection 2023. PMID 37456802